CLINICAL TRIAL: NCT06926231
Title: Impact of a Non-medicinal Technique Medical Hypnosis on Perceived Dyspnea in Difficult Ventilatory Weaning Patients: a Multicenter Randomized Controlled Trial.
Brief Title: Non-medicinal Technique and Dyspnea in Weaning Patients
Acronym: Easy Wean
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 69HCL24_0209; ID-RCB (Other: 2024-A02479-38)
Record Dates: First submitted 2025-03-19; First posted 2025-04-13 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-04

CONDITIONS: Difficult Mechanical Ventilation Weaning; Spontaneous Breathing Trial; Dyspnea
Keywords: difficult mechanical ventilation weaning; dyspnea; mechanical ventilation; spontaneous breathing trial; hypnosis
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medical hypnosis (Experimental): Patients who will receive protocolized medical hypnosis before the SBT every day between inclusion and day-7. Medical hypnosis sessions will consist in the administration of a 5-min hypnotic text by a loudspeaker installed in the ICU room, after selection of a hypnotic theme (sea, mountain or animals) by the participant. The hypnosis session will involve an induction phase, a suggestion phase and an emergence phase, along with self-hypnosis tips. The hypnosis session will immediately precede the SBT (<2h). The intervention is administered before the SBT daily from the randomization to day 7 or until extubation.
  Interventions: Behavioral: Protocolized medical hypnosis
- Standard of care (Active Comparator): Patients who will receive protocolized standard of care (without medical hypnosis) before the SBT, every day between inclusion and day 7.
  Interventions: Behavioral: Protocolized standard of care

INTERVENTIONS:
Behavioral: Protocolized medical hypnosis — Patients who will receive protocolized medical hypnosis before the SBT every day between inclusion and day 7. Medical hypnosis sessions will consist in the administration of a 5-min hypnotic text by a loudspeaker installed in the ICU room, after selection of a hypnotic theme (sea, mountain or animals) by the participant. The hypnosis session will involve an induction phase, a suggestion phase and an emergence phase, along with self-hypnosis tips. The hypnosis session will immediately precede the SBT (<2h). The intervention is administered before the SBT daily from the randomization to day 7 or until extubation.
  Arms: Medical hypnosis
Behavioral: Protocolized standard of care — The protocolized standard of care will consist in the description of authorized human/behavioral patient-nurse interactions and patient installation prior to the daily SBT.
  Arms: Standard of care

SUMMARY:
This is a randomized, controlled, multicenter, open-label, category 2, parallel-arm study of efficacy and superiority.

The target population are patients hospitalized in the intensive care unit (ICU), ventilated with invasive mechanical ventilation for 24 hours or more and having failed a spontaneous breathing trial (SBT, i.e. weaning test of invasive mechanical ventilation [IMV]).

The primary objective is to evaluate the efficacy of medical hypnosis in reducing dyspnea experienced before the SBT in patients identified as difficult to wean in the ICU, compared with the protocolized standard of care.

The primary outcome is the mean value of the daily visual analog scale (VAS) of dyspnea, self-assessed by the patient, measured immediately after the hypnosis session (before SBT) from Day-0 to Day-7 or until extubation. In the control group, the daily value (from D0 to D7 or extubation) of the self-assessed dyspnea VAS will be measured immediately before SBT.

The protocol will be divided into two arms: a control arm in which standard of care practices regarding the daily SBT will be protocolized, and an interventional arm in which patients will receive protocolized medical hypnosis before the daily SBT in addition to the protocolized standard of care. The intervention (hypnosis or control) will be performed daily for 7 days (or until extubation, if applicable). The primary outcome will be assessed daily over the same period.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* hospitalized in the intensive care unit
* receiving invasive mechanical ventilation for 24 hours or more.
* who has failed at least one spontaneous breathing trial

Exclusion Criteria:

* Patient already intubated during current ICU stay (including transfer from another ICU unit), with successful extubation during stay.
* Tracheostomized patient or patient with a short-term tracheostomy project.
* Patients with chronic neuromuscular pathologies (myopathy, amyotrophic lateral sclerosis, multi-system atrophy, non-exhaustive list).
* Patient no longer eligible for SBT at time of inclusion (hemodynamic, neurological or respiratory criterion)
* Psychiatric pathology identified in the medical record, diagnosed by a psychiatrist and for which medication is prescribed (bipolar disorder, schizophrenia, anxiety-depressive disorder, non-exhaustive list).
* Recent brain injury, within < 3 months (stroke, cardiopulmonary arrest with neurological prognosis, non-exhaustive list) objectivated by medical imagery.
* Cognitive impairment or delirium associated with resuscitation, identified by a positive CAM-ICU (Confusion Assessment Method for the Intensive Care Unit) test (dynamic parameter).
* Ocular Glasgow score lower than 4/4 and motor response lower than response to simple commands.
* Delirium tremens with Cushman score > 7 (dynamic parameter).
* Language barrier, patient who does not use French in everyday life.
* Deaf or hearing-impaired patients.
* Re-sedated patient following the failed SBT the day before inclusion.
* Pregnant, parturient or breastfeeding women, objectified by a negative pregnancy test in women of childbearing age.
* Patient for whom a limitation of therapeutics has been decided, including the absence of a re-intubation project.
* Patient whose consent cannot be obtained (directly or in front of a relative or witness).
* Patient already included in the same study or in another study sharing the same primary outcome.
* Patient deprived of liberty by judicial or administrative decision.
* Patient of legal age under legal protection (guardianship, curators).
* Patient not affiliated to a social security system or beneficiary of a similar system.
* Patient participating in another interventional research study with an exclusion period still in effect at pre-inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Mean value of self-reported daily visual analog scale of dyspnea after the intervention or the control strategy | Immediately after the hypnosis session (before SBT) from day 0 to day 7 or until extubation. In the control group, the daily value (from day 0 to day 7 or extubation) of self-reported VAS of dyspnea will be measured immediately before SBT.
  Mean value of self-reported daily visual analog scale (VAS) of dyspnea, measured immediately after the hypnosis session (before SBT) from day 0 to day 7 or until extubation. In the control group, the daily value (from day 0 to day 7 or extubation) of self-reported VAS of dyspnea will be measured immediately before SBT. The outcome measure consists in the mean value of the daily measures collected during this period.

SECONDARY OUTCOMES:
Mean MV-RDOS score (Mechanical Ventilation-Respiratory Distress Observation Scale) after the intervention or the control strategy | Immediately after the hypnosis session (before SBT) from day 0 to day 7 or until extubation. In the control group, the daily value (from day 0 to day 7 or extubation) of MV-RDOS will be measured immediately before SBT.
  The outcome is a scale evaluating respiratory distress assessed by the treating team, as a reliable surrogate of self-reported dyspnea in non-communicative intubated patients The minimum and maximum values are 0 and 16. An RDOS score of less than 3 indicates respiratory comfort; An RDOS score greater than or equal to 3 signifies respiratory distress and need for palliation Higher RDOS scores signify a worsening condition The outcome measure consists in the mean value of the daily measures collected during this period.
Mean VAS of dyspnea at the end of the SBT | Immediately at the end of the daily protocolized SBT, which is performed every day from day 0 to day 7 or until extubation in all patients. Measured daily at the end of the SBT, from day 0 to day 7 or until extubation. Up to 28 days
  Mean value of self-reported daily visual analog scale (VAS) of dyspnea, measured immediately after the hypnosis session (before SBT) from day 0 to day 7 or until extubation. In the control group, the daily value (from day 0 to day 7 or extubation) of self-reported VAS of dyspnea will be measured immediately before SBT.
  The SBT protocol lasts 30 minutes at the end of which the dyspnea VAS will be evaluated.
  The outcome measure consists in the mean value of the daily measures collected during this period.
Mean MV-RDOS at the end of SBT | Immediately at the end of the daily protocolized SBT, which is performed every day from day 0 to day 7 or until extubation in all patients.
  The outcome is a scale evaluating respiratory distress assessed by the treating team, as a reliable surrogate of self-reported dyspnea in non-communicative intubated patients The minimum and maximum values are 0 and 16. An RDOS score of less than 3 indicates respiratory comfort; An RDOS score greater than or equal to 3 signifies respiratory distress and need for palliation Higher RDOS scores signify a worsening condition The SBT protocol lasts 30 minutes at the end of which the MV-RDOS will be evaluated.
  The outcome measure consists in the mean value of the daily measures collected during this period.
Mean VAS of anxiety at the end of SBT | Immediately at the end of the daily protocolized SBT, which is performed every day from day 0 to day 7 or until extubation in all patients.
  Mean value of self-reported daily visual analog scale (VAS) of anxiety, measured immediately after the hypnosis session (before SBT) from day 0 to day 7 or until extubation. In the control group, the daily value (from day 0 to day 7 or extubation) of self-reported VAS of anxiety will be measured immediately before SBT.
  The SBT protocol lasts 30 minutes at the end of which the anxiety VAS will be evaluated. The outcome measure consists in the mean value of the daily measures collected during this period.
Mean VAS of pain at the end of SBT | Immediately at the end of the daily protocolized SBT, which is performed every day from Day 0 to Day 7 or until extubation in all patients. The outcome measure consists in the mean value of the daily measures collected during this period.
  Mean value of self-reported daily visual analog scale (VAS) of pain, measured immediately after the hypnosis session (before SBT) from day 0 to day 7 or until extubation. In the control group, the daily value (from day 0 to day 7 or extubation) of self-reported VAS of pain will be measured immediately before SBT.
  The SBT protocol lasts 30 minutes at the end of which the pain VAS will be evaluated.
Respiratory physiology | Value of respiratory rate and SpO2, measured immediately at the beginning of the SBT, and worst value observed during the daily SBT, between inclusion and day 7 or extubation
  Respiratory rate (in bpm, beats per minute) and O2 percutaneous saturation (in %)
Hemodynamic status | Value of heart rate and mean arterial pressure, measured immediately at the beginning of the SBT, and worst value observed during the daily SBT, between inclusion and day 7 or extubation
  Heart rate (in bpm) and mean arterial pressure (in mmHg / millimetre of mercury)
Quality of applied intervention and control strategies | Up to Day 7
  Rate of medical hypnosis sessions and standard of care sessions in each group achieving predefined quality criteria. Predefined quality criteria are: interruption, quality of the interaction, duration of the intervention, impossibility to apply the strategy, adverse event
Feasibility: enrolment | At the end of the study recruitment.
  Number of subjects included divided by total number of eligible subjects
Feasibility: hypnosis training | At the end of the recruitment.
  Number of hypnosis training sessions for paramedics of participating centers actually carried out in participating centers during the study.
Safety: neurological impact of strategies | The RASS value will be assessed continuously during the duration of the intervention in Gp1 or during the protocolized observation period in Gp2, and its highest value will be reported. It will be reported daily in each group, between inclusion and D7.
  Highest value of the Richmond Agitation Sedation Scale (-5 to +4) observed daily during the hypnosis session or control intervention.
Invasive mechanical ventilation weaning | Measured at day 28
  Ventilator free days (VFD) : number of days alive without invasive mechanical ventilation, between the date of last successful extubation and day 28. A score of 0 is allocated in case of death between inclusion and day 28.
Reintubation | Measured at day 28
  Rate of reintubation within 7 days of extubation, until day 28.
ICU length of stay | through study completion, up to 28 days
  Number of days between randomization and ICU discharge.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Hôpital de Fleyriat - Centre hospitalier de Bourg-en-Bresse - Réanimation Soins continus, Bourg-en-Bresse
  - CHU Clermont Ferrand - Hôpital Gabriel Montpied - Médecine Intensive Réanimation, Clermont-Ferrand
  - CHU Grenoble Alpes - Hôpital Michallon - Médecine Intensive Réanimation, La Tronche
  - Hospices Civils de Lyon - Hôpital de la Croix Rousse - Médecine Intensive Réanimation, Lyon
  - Hospices Civils de Lyon - Hôpital Lyon Sud - Réanimation Polyvalente, Pierre-Bénite